CLINICAL TRIAL: NCT04502862
Title: A Phase 4, Randomized, Double-blind, Placebo-controlled, Multicenter, Parallel-group Study of the Effect of Dupilumab on Sleep Disturbance in Patients With Uncontrolled Persistent Asthma
Acronym: MORPHEO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LPS16677; U1111-1249-6054 (Registry Identifier: ICTRP); 2020-001217-20 (EudraCT Number)
Record Dates: First submitted 2020-08-04; First posted 2020-08-06 (Actual); Results first posted 2024-11-26 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — dupilumab

STUDY DESIGN:
Intervention Model Description: Interim analysis for sample size re-estimation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dupilumab (Experimental): Participants received a loading dose of 400 mg of dupilumab (2 injections × 200 mg) SC on Day 1, followed by 200 mg Q2W for 12 weeks.
  Interventions: Drug: SAR231893
- Placebo (Placebo Comparator): Participants received an initial loading dose of matching placebo (2 injections of placebo) SC on Day 1, followed by 1 injection of placebo Q2W for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SAR231893 — Pharmaceutical form: Solution for injection; Route of administration: Subcutaneous
  Other Names: Dupixent
  Arms: Dupilumab
Drug: Placebo — Pharmaceutical form: Solution for injection; Route of administration: Subcutaneous
  Arms: Placebo

SUMMARY:
Primary Objective:

To assess the effect of dupilumab on sleep

Secondary Objectives:

* To evaluate the effect of dupilumab on additional participant reported sleep outcomes
* To evaluate the effect of dupilumab on objective sleep assessment
* To evaluate the effect of dupilumab on asthma symptoms
* To evaluate the effect of dupilumab on lung function
* To evaluate the safety of dupilumab

DETAILED DESCRIPTION:
Study duration per participant was approximately 16 weeks and up to 29 weeks including up to 5 weeks screening period, a 12-week treatment period and up to 12 weeks post-treatment follow-up period or until the participant switched to commercialized dupilumab (or other biologic product), whichever came first.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of asthma based on the Global Initiative for Asthma (GINA) 2020 Guidelines for ≥12 months treated with medium to high dose inhaled corticosteroid (ICS) and a second controller (ie, long-acting beta agonist, leukotriene receptor antagonist). A third controller is allowed but not mandatory. The dose regimen should be stable for at least 1 month before the study and during the screening period
* History of at least one severe asthma exacerbation within 1 year prior to screening. Severe exacerbation is defined as deterioration of asthma that results in emergency treatment, hospitalization due to asthma, or treatment with systemic steroids (oral or injectable)
* Eosinophils ≥150 cells/μL and fractional exhaled nitric oxide (FeNO) ≥25 ppb during screening, prior to randomization

  * NOTES:
  * Historical values of blood eosinophil count meeting the eligibility criterion measured within 6 months prior to screening Visit 1 in the absence of oral corticosteroid (OCS) treatment are allowed
  * FeNO value to be checked for eligibility at Visit 2 as well
* Asthma control questionnaire (ACQ)-5 ≥2.5 at screening Visit 1 and Visit 2, prior to randomization
* Pre-bronchodilator Forced Expiratory Volume in 1 Second (FEV1) ≤ 80% of predicted normal during screening and at Visit 2, prior to randomization
* Exhibit bronchodilator reversibility (≥12% and 200 mL improvement in FEV1 post short-acting beta agonist administration) during screening period, prior to randomization, unless reversibility test meeting the inclusion criteria was done within 6 months prior to screening Visit 1
* Weekly average nocturnal awakenings due to asthma symptoms in the week prior to screening Visit 1 is ≥1

Exclusion Criteria:

* Current smoker
* Former smoker for 10 years with a smoking history of >10 pack-years
* Severe asthma exacerbation during screening, prior to randomization
* History or clinical evidence of chronic obstructive pulmonary disease (COPD) including Asthma-COPD Overlap Syndrome (ACOS) or any other significant lung disease (eg, lung fibrosis, sarcoidosis, interstitial lung disease, pulmonary hypertension, bronchiectasis, Churg-Strauss Syndrome)
* History of or current evidence of clinically significant non-respiratory diseases that in the opinion of the investigator may interfere with the aims of the study or put the participant at undue risk
* Active tuberculosis (TB) or non-tuberculous mycobacterial infection, or a history of incompletely treated TB will be excluded unless it is well documented by a specialist that the participant has been adequately treated and can now start treatment with a biologic agent, in the medical judgment of the Investigator and/or infectious disease specialist. Tuberculosis testing would be performed on a country by country basis, according to local guidelines if required by Regulatory Authorities or ethics boards
* Diagnosed active endoparasitic infection; suspected or high risk of endoparasitic infection, unless clinical and (if necessary) laboratory assessment have ruled out active infection before randomization
* History of human immunodeficiency (HIV) infection or positive HIV test at screening Visit 1
* Active chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiprotozoals, or antifungals within 2 weeks before screening
* Known or suspected immunodeficiency including history of invasive opportunistic infections, despite infection resolution
* Current evidence of clinically significant oncological disease
* History of systemic hypersensitivity or anaphylaxis to any biologic therapy
* Severe uncontrolled depression
* Sleep disturbances not related to asthma, including sleep apnea, hypersomnia, or insomnia secondary to chronic pain, atopic dermatitis (AD), COPD or other conditions
* Participant who works night shift (ie, any work between 8 pm and 6 am)
* Erratic sleep habits, as determined by the Investigator
* Restless leg syndrome or periodic limb movement disorder
* Chronic treatment with oral corticosteroid (OCS) for more than 2 weeks before screening Visit 1
* Participant taking sedative, anxiolytic, or hypnotic treatments, including melatonin, within 3 months before randomization
* Participant taking systemic sedative antihistamines (excluding newer generations of antihistamines) or theophylline
* Current treatment with antidepressants, lipophilic beta blockers, clonidine, opioids, or other medications known to interfere with sleep and may confound the study assessments, as determined by the Investigator
* Participant who has taken biologic therapy (including dupilumab)/systemic immunosuppressant to treat inflammatory disease or autoimmune disease (eg, rheumatoid arthritis, inflammatory bowel disease, primary biliary cirrhosis, systemic lupus erythematosus, multiple sclerosis, etc) within 2 months or 5 half-lives before screening Visit 1, whichever is longer
* Treatment with live (attenuated) vaccine within 4 weeks before screening Visit 1

  * NOTE: For participants who have vaccination with live, attenuated vaccines planned during the course of the study (based on national vaccination schedule/local guidelines), it will be determined, after consultation with a physician, whether the administration of vaccine can be postponed until after the end of the study, (i.e. after the 12 week follow-up period off-treatment or until the participant switches to commercialized dupilumab or other biologic product, whichever comes first), or preponed to before the start of the study without compromising the health of the participant:
  * Participant for whom administration of live (attenuated) vaccine can be safely postponed would be eligible to enroll into the study
  * Participant who have their vaccination preponed can enroll in the study only after a gap of 4 weeks following administration of the vaccine

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2023-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (55):
- United States (12):
  - Kern Allergy and Medical Research. Inc. Site Number : 8400003, Bakersfield, California
  - Todd Astor MD Site Number : 8400016, Culver City, California
  - Southern California Institute for Respiratory Diseases Site Number : 8400009, Los Angeles, California
  - Allergy & Asthma Associates of Santa Clara Valley Site Number : 8400001, San Jose, California
  - Asthma and Allergy Associates, PC Site Number : 8400011, Colorado Springs, Colorado
  - Sarasota Clinical Research Site Number : 8400012, Sarasota, Florida
  - Allergy & Asthma Specialists, PSC Site Number : 8400004, Owensboro, Kentucky
  - The Asthma and Allergy Center Site Number : 8400010, Bellevue, Nebraska
  - OK Clinical Research LLC Site Number : 8400005, Edmond, Oklahoma
  - Velocity Clinical Research, Medford Site Number : 8400007, Medford, Oregon
  - National Allergy and Asthma Research, LLC Site Number : 8400008, Charleston, South Carolina
  - TTS Research Site Number : 8400006, Boerne, Texas
- Argentina (5):
  - Investigational Site Number : 0320003, CABA, Buenos Aires
  - Investigational Site Number : 0320001, CABA, Buenos Aires
  - Investigational Site Number : 0320004, Rosario, Santa Fe Province
  - Investigational Site Number : 0320005, Rosario, Santa Fe Province
  - Investigational Site Number : 0320002, Buenos Aires
- Canada (4):
  - Investigational Site Number : 1240012, Ajax, Ontario
  - Investigational Site Number : 1240005, Toronto, Ontario
  - Investigational Site Number : 1240009, Québec
  - Investigational Site Number : 1240008, Windsor
- Germany (6):
  - Investigational Site Number : 2760002, Berlin
  - Investigational Site Number : 2760005, Frankfurt am Main
  - Investigational Site Number : 2760003, Hanover
  - Investigational Site Number : 2760001, Koblenz
  - Investigational Site Number : 2760004, Leipzig
  - Investigational Site Number : 2760006, Lübeck
- Italy (3):
  - Investigational Site Number : 3800006, Monserrato, Cagliari
  - Investigational Site Number : 3800001, Orbassano, Torino
  - Investigational Site Number : 3800005, Reggio Emilia
- Netherlands (3):
  - Investigational Site Number : 5280005, Arnhem
  - Investigational Site Number : 5280001, Breda
  - Investigational Site Number : 5280002, Leeuwarden
- Portugal (5):
  - Investigational Site Number : 6200001, Aveiro
  - Investigational Site Number : 6200007, Guimarães
  - Investigational Site Number : 6200006, Lisbon
  - Investigational Site Number : 6200003, Matosinhos Municipality
  - Investigational Site Number : 6200004, Porto
- Russia (6):
  - Investigational Site Number : 6430001, Moscow
  - Investigational Site Number : 6430002, Moscow
  - Investigational Site Number : 6430006, Moscow
  - Investigational Site Number : 6430005, Moscow
  - Investigational Site Number : 6430007, Saint Petersburg
  - Investigational Site Number : 6430004, Saint Petersburg
- Spain (3):
  - Investigational Site Number : 7240001, Lugo / Lugo, Galicia [Galicia]
  - Investigational Site Number : 7240002, Valencia, Valenciana, Comunidad
  - Investigational Site Number : 7240005, Madrid
- Ukraine (6):
  - Investigational Site Number : 8040002, Ivano-Frankivsk
  - Investigational Site Number : 8040006, Ivano-Frankivsk
  - Investigational Site Number : 8040003, Kharkiv
  - Investigational Site Number : 8040008, Kyiv
  - Investigational Site Number : 8040007, Kyiv
  - Investigational Site Number : 8040005, Vinnytsia
- United Kingdom (2):
  - Investigational Site Number : 8260001, Cambridge, Cambridgeshire
  - Investigational Site Number : 8260002, London, London, City of

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: LPS16677 Plain language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25288&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 52 centers in 11 countries. A total of 397 participants were screened between 10 August 2020 to 30 May 2023, of which 195 participants were screen failures. Screen failures were mainly due to not meeting the eligibility criteria.
Pre-assignment Details: A total of 202 participants were randomized in a ratio of 1:1 to receive dupilumab or matching placebo every 2 weeks (Q2W) for 12 weeks.
Groups:
- Dupilumab 200 mg Q2W: Participants received a loading dose of 400 milligrams (mg) of dupilumab (2 injections × 200 mg) subcutaneous (SC) on Day 1, followed by 200 mg Q2W for 12 weeks.
Period: Overall Study
Arm/Group | Dupilumab 200 mg Q2W | Placebo
Started (Randomized) | 101 | 101
Randomized and Treated | 100 | 101
Completed | 95 | 94
Not Completed | 6 | 7
Not completed — Not Related to Coronavirus Disease-2019 (COVID-19) pandemic | 4 | 6
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat (ITT) analysis set consisted of all randomized participants.
Groups:
- Dupilumab 200 mg Q2W: Participants received a loading dose of 400 mg of dupilumab (2 injections × 200 mg) SC on Day 1, followed by 200 mg Q2W for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Dupilumab 200 mg Q2W | Placebo | Total
Number analyzed (Participants) | 101 | 101 | 202
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.9 (12.63) | 46.6 (12.71) | 46.7 (12.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 76 | 144
  Male | 33 | 25 | 58
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 4 | 4 | 8
  White | 92 | 92 | 184
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1
Sleep Disturbance Score [Mean (Standard Deviation); unit: Score on a scale] — Sleep disturbance score was assessed by Asthma Sleep Disturbance Questionnaire (ASDQ). Participants recorded severity of disturbance of sleep due to asthma as: 0 = slept through night, no asthma symptoms; 1 = slept well, no night time awakenings because of asthma, but some asthma symptoms in the morning; 2 = woke up once because of asthma; 3 = woke up several times because of asthma and 4 = bad night, awake most of the night because of asthma. Total scores ranges between 0 (no impact of asthma on sleep) and 4 (higher impact of asthma on sleep). Higher scores indicated worse outcomes. Population: Only those participants with data available at baseline are reported.
  Score on a scale
    number analyzed (Participants) | 99 | 98 | 197
    (all) | 1.89 (0.769) | 1.83 (0.754) | 1.86 (0.760)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in Sleep Disturbance Score Using the Asthma Sleep Disturbance Questionnaire (ASDQ)
Description: The ASDQ is a participant-reported outcome (PRO) measure designed to assess the impact of asthma on participants' sleep. Participants were instructed to record the severity of the disturbance of their sleep due to asthma as: 0 = slept through the night, no asthma symptoms; 1 = slept well, no night time awakenings because of asthma, but some asthma symptoms in the morning; 2 = woke up once because of asthma (may or may not include early awakening); 3 = woke up several times because of asthma (may or may not include early awakening) and 4 = bad night, awake most of the night because of asthma. The participants recorded their sleep disturbance in an electronic diary, once a day upon awakening. Total scores ranges between 0 to 4 with 0 indicating no impact of asthma on sleep and 4 indicating higher impact of asthma on sleep. Higher scores indicated worse outcomes. Baseline was calculated by averaging the data collected/recorded from Day -6 to Day 1.
Time Frame: Baseline (Day -6 to Day 1) up to Week 12
Population: The ITT for primary endpoint (ITTp) analysis set consisted of all ITT participants excluding those who used the original version of sleep disturbance questionnaire at baseline and/or post-baseline included in the mixed effect model for repeated measures (MMRM) model. Only those participants with data collected at baseline and at least one post-baseline until Week 12 are reported.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Dupilumab 200 mg Q2W | Placebo
Number analyzed (Participants) | 94 | 93
Score on a scale | -0.88 (0.077) | -0.81 (0.077)
Statistical Analysis 1: Comparison: Dupilumab 200 mg Q2W vs Placebo; The MMRM model included study intervention, age, body mass index (BMI), region (Eastern Europe, rest of world [ROW]), inhaled corticosteroids [ICS] dose level at baseline (ICS dose level medium, ICS dose level high), visit (up to Week 12), study intervention-by-visit interaction, baseline asthma control questionnaire (ACQ-5), baseline sleep disturbance score and baseline-by-visit interaction as covariates; Test type: Other; p = 0.512, MMRM — A hierarchical testing procedure was used to control type I error and handle primary and first 2 secondary endpoints (reported sequentially) analyses at a 2-sided significance level of 0.05; Least square mean difference = -0.07, 95% CI 2-sided [-0.28 to 0.14], Standard Error of Mean 0.107

2. Secondary Outcome: Change From Baseline to Week 12 on the Number of Nocturnal Awakenings (Sleep Diary)
Description: Sleep diary is used to assess adult sleep disturbance due to asthma. Number of nocturnal awakenings was determined based on answer on question from sleep diary: "Approximately how many times did you wake up last night (not including when you woke up for the day today)?" Baseline was calculated by averaging the data collected/recorded from Day -6 to Day 1.
Time Frame: Baseline (Day -6 to Day 1) up to Week 12
Population: The ITT analysis set consisted of all randomized participants included in the MMRM model. Only those participants with data collected at baseline and at least one post-baseline until Week 12 are reported.
Measure: Least Squares Mean (Standard Error); unit: Number of nocturnal awakenings
Arm/Group | Dupilumab 200 mg Q2W | Placebo
Number analyzed (Participants) | 98 | 98
Number of nocturnal awakenings | -0.71 (0.080) | -0.71 (0.080)
Statistical Analysis 1: Comparison: Dupilumab 200 mg Q2W vs Placebo; The MMRM model included study intervention, age, BMI, region (Eastern Europe, ROW), ICS dose level at baseline (ICS dose level medium, ICS dose level high), visit (up to Week 12), study intervention-by-visit interaction, baseline ACQ-5, baseline number of nocturnal awakenings and baseline-by-visit interaction as covariates; Test type: Other; p = 0.967, MMRM — [p-value comment as in outcome 1, analysis 1]; Least square mean difference = 0.00, 95% CI 2-sided [-0.21 to 0.22], Standard Error of Mean 0.110

3. Secondary Outcome: Change From Baseline to Week 12 in Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep-Related Impairment 8a Scale
Description: PROMIS sleep-related impairment eight-term 8a scale was administered to assess impact of sleep-related impairment during waking hours. The questionnaire focuses on self-reported perceptions of alertness, sleepiness, and tiredness during usual waking hours, and perceived functional impairments during wakefulness associated with sleep problems or impaired alertness. It assesses sleep-related impairment over the past 7 days. Each item is rated on a 5-point scale (1 = not at all; 2 = a little bit; 3 = somewhat; 4 = quite a bit; and 5 = very much) with a raw score from 8 to 40 with higher scores indicating greater sleep impairment. PROMIS T-score is presented which rescales the raw score into a standardized score with a mean of 50 and a standard deviation of 10. Possible range for T-score=30 to 80; higher scores=greater severity of sleep impairment. Baseline=last available valid (non-missing) value up to and including the day of first dose of investigational medicinal product (IMP).
Time Frame: Baseline (Day 1) up to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Dupilumab 200 mg Q2W | Placebo
Number analyzed (Participants) | 97 | 96
T-score | -7.20 (0.624) | -6.51 (0.626)
Statistical Analysis 1: Comparison: Dupilumab 200 mg Q2W vs Placebo; The MMRM model included study intervention, age, BMI, region (Eastern Europe, ROW), ICS dose level at baseline (ICS dose level medium, ICS dose level high), visit (up to Week 12), study intervention-by-visit interaction, baseline ACQ-5, baseline PROMIS total score and baseline-by-visit interaction as covariates; Test type: Other; p = 0.422, MMRM — [p-value comment as in outcome 1, analysis 1]; Least square mean difference = -0.70, 95% CI 2-sided [-2.40 to 1.01], Standard Error of Mean 0.865

4. Secondary Outcome: Change From Baseline to Week 12 in Sleep Quality (Sleep Diary)
Description: Sleep diary is used to assess adult sleep disturbance due to asthma. Sleep quality was assessed on a 11-point scale which ranged from 0 (worst possible sleep) to 10 (best possible sleep); higher scores indicated better outcomes. Baseline was calculated by averaging the data collected/recorded from Day -6 to Day 1.
Time Frame: Baseline (Day -6 to Day 1) up to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Dupilumab 200 mg Q2W | Placebo
Number analyzed (Participants) | 98 | 98
Score on a scale | 1.14 (0.151) | 0.97 (0.152)

5. Secondary Outcome: Change From Baseline to Week 12 in Restorative Sleep (Sleep Diary)
Description: Sleep Diary is used to assess adult sleep disturbance due to asthma. Question about restorative sleep asks participants to recall "when they got up for the day today". Restorative sleep was assessed on a 11-point scale which ranged from 0 (worst possible sleep) to 10 (best possible sleep); higher scores indicated better outcomes. Baseline was calculated by averaging the data collected/recorded from Day -6 to Day 1.
Time Frame: Baseline (Day -6 to Day 1) up to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Dupilumab 200 mg Q2W | Placebo
Number analyzed (Participants) | 98 | 98
Score on a scale | 1.15 (0.152) | 1.02 (0.152)

6. Secondary Outcome: Change From Baseline to Week 12 in Wake After Sleep Onset (WASO) (Sleep Diary)
Description: Sleep Diary is used to assess adult sleep disturbance due to asthma. WASO was calculated as time awake after initial sleep onset but before the final awakening. Baseline was calculated by averaging the data collected/recorded from Day -6 to Day 1.
Time Frame: Baseline (Day -6 to Day 1) up to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Dupilumab 200 mg Q2W | Placebo
Number analyzed (Participants) | 98 | 98
Minutes | -30.58 (3.945) | -26.48 (3.962)

7. Secondary Outcome: Change From Baseline to Week 12 in WASO Based on Actigraphy Data
Description: Wrist actigraphy is a procedure that records and integrates occurrence and degree of limb movement activity over an extended recording period. The signals generated by wrist movement are sensed by a tiny microcomputer contained within watch and translated into activity counts. Algorithms have been developed to translate these activity counts or "epochs" (or "periods") that correspond to times when a person is likely to be asleep or wake. Actigraph was worn on wrist of non-dominant hand to provide estimates of duration, timing and patterns of sleep in study participants. After the watch data were scored by a selected expert center, a number of summary measurements were generated for each participant, including WASO. Baseline was calculated by averaging the data collected/recorded from Day -6 to Day 1.
Time Frame: Baseline (Day -6 to Day 1) up to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Dupilumab 200 mg Q2W | Placebo
Number analyzed (Participants) | 84 | 92
Minutes | -1.64 (2.286) | -1.17 (2.215)

8. Secondary Outcome: Change From Baseline to Week 12 in Asthma Daytime Symptom Diary (ADSD)
Description: The ADSD is a PRO measure designed to measure asthma symptoms in adult and adolescent (12 years of age and older) participants diagnosed with mild to severe asthma. ADSD assesses asthma severity based on participant self-report of asthma core symptoms, i.e., difficulty breathing, wheezing, shortness of breath, chest tightness, chest pain, and cough. Participants were asked to complete the ADSD every night before they go to bed, thinking about their asthma symptoms today, from when they got up this morning until now. ADSD is composed of 6 items rated using an 11-point NRS that ranges from 0 = None to 10 = as bad as you can imagine. The total score was calculated by averaging all 6 items and therefore the score ranged from 0 to 10. Higher scores indicated worse outcomes. Baseline value was average of the data from Day -7 to Day -1.
Time Frame: Baseline (Day -7 to Day -1) up to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Dupilumab 200 mg Q2W | Placebo
Number analyzed (Participants) | 71 | 70
Score on a scale | -1.78 (0.192) | -1.56 (0.193)

9. Secondary Outcome: Change From Baseline to Week 12 in Asthma Nighttime Symptom Diary (ANSD)
Description: The ANSD is a PRO measure designed to measure asthma symptoms in adult and adolescent (12 years of age and older) participants diagnosed with mild to severe asthma. ANSD assesses asthma severity based on participant self-report of asthma core symptoms, i.e., difficulty breathing, wheezing, shortness of breath, chest tightness, chest pain, and cough. Participants were asked to complete the ANSD when getting up, thinking about their asthma symptoms last night from when they went to bed until now. ANSD is composed of 6 items rated using an 11-point NRS that ranges from 0 = None to 10 = as bad as you can imagine. The total score was calculated by averaging all 6 items and therefore the score ranged from 0 to 10. Higher scores indicated worse outcomes. Baseline value was average of the data from Day -6 to Day -1.
Time Frame: Baseline (Day -6 to Day -1) up to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Dupilumab 200 mg Q2W | Placebo
Number analyzed (Participants) | 85 | 85
Score on a scale | -1.58 (0.178) | -1.36 (0.178)

10. Secondary Outcome: Change From Baseline to Week 12 in Pre-Bronchodilator Forced Expiratory Volume (Pre-BD FEV1)
Description: FEV1 was the volume of air exhaled in the first second of a forced expiration as measured by spirometer. For pre-BD FEV1, spirometry was performed before IMP administration and after withholding the standard of care asthma treatment which was verified before performing the measurements. Baseline was defined as the last available valid (non-missing) value up to and including the day of first dose of IMP.
Time Frame: Baseline (Day 1) up to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Dupilumab 200 mg Q2W | Placebo
Number analyzed (Participants) | 100 | 99
Liter | 0.49 (0.044) | 0.27 (0.047)

11. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Treatment-Emergent Serious Adverse Events (TESAEs), and Treatment-Emergent Adverse Events Of Special Interest (TEAESIs)
Description: AE: any untoward medical occurrence in participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAEs: AEs that developed or worsened or became serious during TEAE period, defined as time from first administration of IMP (on Day 1) to last administration of IMP + 98 days or until participant switches to commercialized dupilumab or other biologics. SAE: any untoward medical occurrence that, at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. AESI: AE (serious or nonserious) of scientific and medical concern specific to Sponsor's product or program, for which ongoing monitoring and immediate notification by Investigator to Sponsor is required.
Time Frame: From first dose of study drug (Day 1) up to 12 weeks after last dose of study drug, approximately 30 weeks
Population: Safety analysis set included all randomized participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Dupilumab 200 mg Q2W | Placebo
Number analyzed (Participants) | 100 | 101
Participants
  Any TEAE | 48 | 46
  Any TESAE | 3 | 3
  Any TEAESI | 0 | 0

12. Secondary Outcome: Number of Participants With Potentially Clinically Significant Abnormalities (PCSA) in Vital Signs
Description: Vital signs included systolic blood pressure (SBP), diastolic blood pressure (DBP), heart rate (HR) and weight. Criteria for PCSA: SBP: ≤95 millimeters of mercury (mmHg) and decrease from baseline ≥20 mmHg, ≥160 mmHg and increase from baseline ≥20 mmHg; DBP: ≤45 mmHg and decrease from baseline ≥10 mmHg, ≥ 110 mmHg and increase from baseline ≥ 10 mmHg; HR: ≤ 50 beats per minute (bpm) and decrease from baseline ≥ 20 bpm, ≥120 bpm and increase from baseline ≥ 20 bpm; Weight: ≥ 5% increase from baseline, ≥5% decrease from baseline.
Time Frame: From first dose of study drug (Day 1) up to 12 weeks after last dose of study drug, approximately 30 weeks
Population: Safety analysis set included all randomized participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Dupilumab 200 mg Q2W | Placebo
Number analyzed (Participants) | 100 | 101
Participants
  SBP: ≤95 mmHg and decrease from baseline ≥20 mmHg | 0 | 1
  SBP: ≥160 mmHg and increase from baseline ≥20 mmHg | 1 | 2
  DBP: ≤45 mmHg and decrease from baseline ≥10 mmHg | 0 | 0
  DBP: ≥ 110 mmHg and increase from baseline ≥ 10mmHg | 0 | 0
  HR: ≤ 50 bpm and decrease from baseline ≥ 20 bpm | 0 | 0
  HR: ≥ 120 bpm and increase from baseline ≥ 20 bpm | 0 | 0
  Weight: ≥5% increase from baseline | 3 | 6
  Weight: ≥5% decrease from baseline | 5 | 4

ADVERSE EVENTS:
Time Frame: TEAEs were collected from first dose of study drug (Day 1) up to 12 weeks after last dose of study drug, approximately 30 weeks. All-cause mortality (deaths) were collected from first dose of study drug (Day 1) up to end of study, approximately 39 months.
Description: Analysis was performed on safety population.
Arm/Group | Dupilumab 200 mg Q2W | Placebo
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/101
Serious Adverse Events (participants affected / at risk) | 3/100 | 3/101
Other Adverse Events (participants affected / at risk) | 13/100 | 18/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dupilumab 200 mg Q2W (N=100) | Placebo (N=101)
Pancreatitis Acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Covid-19 Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Depression Suicidal (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide Attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dupilumab 200 mg Q2W (N=100) | Placebo (N=101)
Nasopharyngitis (Infections and infestations) | 4 (4) | 7 (7)
Asthma (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 14 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2022-09-22): https://cdn.clinicaltrials.gov/large-docs/62/NCT04502862/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-09): https://cdn.clinicaltrials.gov/large-docs/62/NCT04502862/SAP_001.pdf